CLINICAL TRIAL: NCT02616133
Title: HER2+ Breast Cancer Neo-Adjuvant Coordination of Care Program
Acronym: CECity
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00064108
Record Dates: First submitted 2015-11-09; First posted 2015-11-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: chart abstraction — abstraction of breast cancer patients with de-identified data

SUMMARY:
Currently many patients with HER2+ Breast Cancer do not have the opportunity to be evaluated by a medical oncologist for neo-adjuvant treatment due to the current lack of care coordination between the surgeon/surgical oncologist and the medical oncologists.

This project will evaluate the feasibility to enhance knowledge that drives adoption of evidence based care, and evaluate the improvement in care coordination between oncologists and surgeons for patients with HER2+ Breast Cancer in the Neo-Adjuvant setting.

DETAILED DESCRIPTION:
The HER2+ Breast Cancer Neo-Adjuvant Coordination of Care Program will evaluate the feasibility, effectiveness, and adoption of evidence based medicine for patients with HER2+ breast cancer through a care coordination application hosted on CECity's MedConcert™ platform. The goal is to implement evidence into practice using existing patient data, and to improve care based on knowledge that will enable care coordination between medical oncologists and surgeons.

PHASE 1: Workflow Design The steering committee from Duke has created a workflow process related to the HER2+ Neo-Adjuvant Therapy Treatment. The goal of the workflow is to establish a coordinated approach to care and identifying key steps in the process. The workflow will identify if the patient had a timely engagement of the multidisciplinary team; if a pre-treatment assessment was performed; if neo-adjuvant therapy treatment was prescribed; if appropriate management and adherence to treatment as prescribed occurred; if surgery was performed and the identification of the type of surgery; and if any subsequent therapy was prescribed. Data collection will be performed at each of the steps in the workflow.

PHASE 2: Engagement Three sites were identified to participate in the project. Each is affiliated with the Duke Cancer Network and are free standing hospital systems and clinics. A coordinator will be designated at each site to guide the process, enter data and communicate patient progress to the sites multidisciplinary project team. Routine communication will be maintained between each site and the project team to ensure timely resolution of any issues or to answer questions.

PHASE 3: Feedback Performance measures have been identified for which data will be collected and aggregated. The data will be displayed in a performance monitor in the CECity MedConcert™ application to provide feedback to providers on their performance related to the measures. Providers will also be provided access to educational resources and improvement opportunities through the application.

PHASE 4: Assessment of Change and Dissemination of Findings Currently, many patients with HER2+ Breast Cancer do not have the opportunity to be evaluated by an oncologist for neo-adjuvant treatment because of a lack of coordinated care between surgeons and oncologists. This project will evaluate adopting evidence-based medicine for patients with HER2+ through the use of a coordinated care application. The goal is to facilitate greater coordination of care between oncologists and surgeons and to identify interventions for improved care. A final report will outline the results of the coordinated care approach. The results of this QI initiative will be developed into a manuscript for publication.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer

Exclusion Criteria:

* no diagnosis of breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Identified patient with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Coordination of Care efforts evaluation score | 6 months to one year
  Multiple measurements will be aggregated from across study sites to evaluate coordination of care efforts across different disciplines involved in the care of a breast cancer patient.This evaluation will result in the formation of a multidisciplinary approach to care for breast cancer subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Sutton, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Marquette General Hospital, Marquette, Michigan
  - DLP Maria Parham Medical Center, Henderson, North Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Augusta Health, Fishersville, Virginia